CLINICAL TRIAL: NCT04203056
Title: Aripiprazole Lauroxil for Preventing Psychotic Relapse After an Initial Schizophrenia Episode
Acronym: APPRAISE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Withdraw of financial support by industry collaborator
Sponsor: University of California, Los Angeles (Other)
Collaborators: Alkermes, Inc. (Industry)
Responsible Party: Principal Investigator, Kenneth L. Subotnik, PhD, Project Scientist, Adjunct Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PATS 20184225
Record Dates: First submitted 2019-12-16; First posted 2019-12-18 (Actual); Results first posted 2023-11-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Schizophrenia; Schizoaffective Disorder, Depressive Type; Schizophreniform Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — aripiprazole lauroxil; Aripiprazole

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial; 12-month longitudinal follow-through study (anticipate enrolling at least 128 patients of whom 90 will be randomized to one of the two arms)
Masking Description: open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- AL-LAI: Long-Acting Injectable Antipsychotic (Experimental): Patients successfully completing the Stabilization period will be randomized to one of the two medications groups: For patients assigned to the AL-LAI (aripiprazole lauroxil- long-acting injections), initiation of AL-LAI will begin with a one-day initiation regimen (using AL-NCD IM (aripiprazole lauroxil NanoCrystal Dispersion)). Subsequent dosing of AL-LAI will be flexible based on clinician judgment. Treatment with AL-LAI can be initiated at a dose of 441mg or 661mg (administered monthly), 882mg (administered monthly or every 6 weeks), or 1064mg (administered every 2 months). Note: These dosages are not assigned levels of the intervention and dosage levels may be changed at any time throughout the 12-month intervention based on clinical need and clinician judgement. Starting dosages do not indicate separate treatment conditions.
  Interventions: Drug: Aripiprazole Lauroxil; Drug: AL-NCD
- ARI-ORAL: Aripiprazole Oral Antipsychotic (Active Comparator): Patients successfully completing the Stabilization period will be randomized to one of the two medications groups: Patients assigned to the oral medication condition will continue with ARI-ORAL. ARI-ORAL dosage will be flexible and dosage will be at the discretion of the treating psychiatrist. Patients discontinuing ARI-ORAL study drug after Randomization to oral antipsychotic medication, can remain in active treatment and follow-up within the study, and may be prescribed any of a number of first-line oral antipsychotics.
  Interventions: Drug: ARI-ORAL

INTERVENTIONS:
Drug: Aripiprazole Lauroxil — 12 month longitudinal aripiprazole lauroxil treatment and assessment follow-through
  Other Names: Aristada
  Arms: AL-LAI: Long-Acting Injectable Antipsychotic
Drug: ARI-ORAL — oral aripiprazole
  Other Names: aripiprazole; Abilify
  Arms: ARI-ORAL: Aripiprazole Oral Antipsychotic
Drug: AL-NCD — Aripiprazole Lauroxil 675 MG/2.4 ML Intramuscular Suspension, Extended Release
  Other Names: Aristada Initio
  Arms: AL-LAI: Long-Acting Injectable Antipsychotic

SUMMARY:
This 12-month study will evaluate the efficacy of aripiprazole lauroxil compared to oral aripiprazole in preventing the re-emergence of psychotic symptoms in patients with a recent onset of schizophrenia.

DETAILED DESCRIPTION:
This is a single-site 12-month open-label randomized study comparing the efficacy of the FDA-approved long-acting formulation of aripiprazole lauroxil to the efficacy of oral aripiprazole among patients with a recent onset of schizophrenia, schizophreniform, or schizoaffective (depressed) disorder. All assessments and treatment will take place at the UCLA Aftercare Research Program (300 UCLA Medical Plaza, Los Angeles, CA 90095), which is a program that specializes in the treatment and study of individuals with a recent onset of schizophrenia. The primary goal is to evaluate the efficacy of aripiprazole lauroxil compared to oral aripiprazole in preventing the re-emergence of psychotic symptoms in patients with a recent onset of schizophrenia. All patients on oral medications will, at least initially, be treated with oral aripiprazole.

ELIGIBILITY:
Inclusion Criteria:

1. Is between 18 and 45 years of age, inclusive, at Screening.
2. Has a diagnosis of schizophreniform disorder, schizophrenia, or schizoaffective disorder, depressed type.
3. Has a first episode of a psychotic illness that occurred within the 24 months before entry.
4. Fluency (oral and written) in the English language.
5. Exhibits tolerability to ARI ORAL during the Stabilization period.
6. Resides within commuting distance of the UCLA Aftercare Research Program in a stable living situation where the patient can be located.
7. Agrees to abide by the contraceptive requirements of the protocol.
8. Additional criteria may apply

Exclusion Criteria:

1. Evidence of a known neurological disorder (e.g., epilepsy) or significant head injury.
2. Premorbid IQ less than 70.
3. Is currently pregnant or breastfeeding, or is planning to become pregnant during the study.
4. Is currently on a long-acting injectable antipsychotic medication and it is clinically contra-indicated to switch to oral aripiprazole.
5. History of poor or inadequate response to an adequate trial of oral or injectable aripiprazole.
6. Has received AL-LAI or IM depot aripiprazole within two months prior to Randomization.
7. Has alcohol or substance abuse as a prominent clinical problem or makes the primary diagnosis not possible to confirm.
8. Is currently being treated with clozapine.
9. Has participated in a clinical drug trial involving any drug within the past two months.
10. Has a current DSM-5 diagnosis of bipolar disorder, or schizoaffective disorder, bipolar type, based on the screening SCID.
11. Patient is an imminent danger to himself/herself.
12. History of neuroleptic malignant syndrome, malignant hyperthermia, or clinically significant tardive dyskinesia.
13. Additional criteria may apply.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth L Subotnik, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- AL-LAI: Long-Acting Injectable Antipsychotic: Patients successfully completing the Stabilization period will be randomized to one of the two medications groups: For patients assigned to the AL-LAI (aripiprazole lauroxil- long-acting injections), initiation of AL-LAI will begin with a one-day initiation regimen (using AL-NCD IM (aripiprazole lauroxil NanoCrystal Dispersion)). Subsequent dosing of AL-LAI will be flexible based on clinician judgment. Treatment with AL-LAI can be initiated at a dose of 441mg or 661mg (administered monthly), 882mg (administered monthly or every 6 weeks), or 1064mg (administered every 2 months).
  Aripiprazole Lauroxil: 12 month longitudinal aripirprazole lauroxil treatment and assessment follow-through
  AL-NCD: Aripiprazole Lauroxil 675 MG/2.4 ML Intramuscular Suspension, Extended Release
Period: Overall Study
Arm/Group | AL-LAI: Long-Acting Injectable Antipsychotic | ARI-ORAL: Aripiprazole Oral Antipsychotic
Started | 6 | 9
Completed | 3 | 5
Not Completed | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AL-LAI: Long-Acting Injectable Antipsychotic | ARI-ORAL: Aripiprazole Oral Antipsychotic | Total
Number analyzed (Participants) | 6 | 9 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.2 (2.6) | 25.9 (7.3) | 24.5 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 3 | 6 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 2 | 5 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 3 | 3 | 6
  More than one race | 1 | 4 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 9 | 15

OUTCOME MEASURES:

1. Primary Outcome: Exacerbation or Relapse of Psychotic Symptoms
Description: Number of participants who experienced an exacerbation and/or relapse following a period of absence or relative low levels of psychotic symptoms based on the expanded 24-item version of the Brief Psychiatric Rating Scale
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | AL-LAI: Long-Acting Injectable Antipsychotic | ARI-ORAL: Aripiprazole Oral Antipsychotic
Number analyzed (Participants) | 6 | 9
Participants | 2 | 2

2. Secondary Outcome: Change in Role Ratings on the Global Functioning Scale From Baseline to 12 Months
Description: The groups will be compared on change in this measure of role functioning. Scores range from 1 to 10, with higher indicating better role functioning. Change scores can theoretically range from 0 to 9
Time Frame: mean change from baseline to the 12 month point
Population: Fewer subjects analyzed than enrolled because only 6 subjects reached the 12 month point and had role functioning data availabe prior to study discontinuation.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | AL-LAI: Long-Acting Injectable Antipsychotic | ARI-ORAL: Aripiprazole Oral Antipsychotic
Number analyzed (Participants) | 2 | 4
score on a scale | 4.3 (.97) | .06 (.97)

3. Secondary Outcome: Change From Baseline to One-Year in the "MATRICS Consensus Cognitive Battery (MCCB)" Overall Composite T-Score.
Description: The change from Baseline to One-year on the MATRICS Consensus Cognitive Battery Overall Composite score. MATRICS is the abbreviation for Measurement and Treatment Research to Improve Cognition in Schizophrenia. T scores do not have an absolute minimum or maximum. Higher scores represent better cognition. The sex and age adjusted T-score was used. The T-Score has a population mean of 50 and standard deviation of 10.
  Fewer subjects analyzed than enrolled because only 9 subjects reached the 12 month point by study discontinuation and had MCCB data.
Time Frame: 12 months
Measure: Mean (Standard Error); unit: Change score: change in T scores
Arm/Group | AL-LAI: Long-Acting Injectable Antipsychotic | ARI-ORAL: Aripiprazole Oral Antipsychotic
Number analyzed (Participants) | 4 | 5
Change score: change in T scores | 9.3 (2.2) | 4.6 (2.5)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time of enrollment (signing the informed consent form) until completing the 12 month protocol or withdrawing early.
Description: Note: Dosages are not assigned levels of the intervention and dosage levels may be changed at any time throughout the 12-month intervention based on clinical need and clinician judgement. Starting dosages do not indicate separate treatment conditions. Therefore, Adverse events are not separated according to starting dosage. In any case, there were no serious adverse events to report for patients in the AL-LAI arm of the study.
Arm/Group | AL-LAI: Long-Acting Injectable Antipsychotic | ARI-ORAL: Aripiprazole Oral Antipsychotic
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/9
Other Adverse Events (participants affected / at risk) | 0/6 | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AL-LAI: Long-Acting Injectable Antipsychotic (N=6) | ARI-ORAL: Aripiprazole Oral Antipsychotic (N=9)
Arrest (Psychiatric disorders) | 0 (0) | 1 (1) — Arrested following property damage while psychotic and nonadherent with aripiprazole.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-07): https://cdn.clinicaltrials.gov/large-docs/56/NCT04203056/Prot_SAP_001.pdf